CLINICAL TRIAL: NCT06720103
Title: Correlation Between Radiculopathy And Quality Of Life In Patients With Chronic Lumbar Spondylosis
Acronym: LS
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Abdelmageed Ali, principale investigator: mona abdelmageed ali, Cairo University
Other Study IDs: P.T.REC/012/005463
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Lumbar Spondylosis
Keywords: quality of life; radiculopathy; lumbar spondylosis
MeSH Terms: conditions — Spondylosis; Radiculopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lumbar spondylosis patients: one hundred thirty-two subjects (who have chronic lumbar spondylosis); from both genders will participate in this group.

SUMMARY:
This study will be conducted to answer the following question:

Is there a Correlation Between Lumbar Radiculopathy and Quality of Life in Patients with chronic lumbar spondylosis?

DETAILED DESCRIPTION:
Spondylosis is an age-related change of vertebrae and discs of the spine. These changes are often called degenerative disc disease and osteoarthritis. When this condition is in the lower back, it's called lumbar spondylosis.

Lumbar osteoarthritis, disc degeneration, degenerative disc disease, and spondylosis are some of the terms used to describe disc changes. In fact, the condition is called spondylosis. Whenever there is a degeneration co-occurrence in the disc, the lumbar spine, the formation of osteophytes and the associated changes in the nerves and the resulting symptoms of pain.Spinal osteoarthritis (OA) is a degenerative process defined radiologically by joint space narrowing, osteophytosis, subchondral sclerosis, and cyst formation.

Osteophytes included within this definition fall into one of the two primary clinical categories.

The first, spondylosis deforms describes bony outgrowths arising primarily along the anterior and lateral perimeters of the vertebral endplate apophyses. These hypertrophic changes are believed to develop at sites of stress to the annular ligament and most commonly occur at thoracic T9-10 and lumbar L3 levels.These conditions lead to nerve root compression, resulting in radiating pain down the leg, commonly referred to as sciatica. The impact of lumbar radiculopathy extends beyond pain, affecting muscle function and neuromuscular control. The involvement of nerve roots such as L4, L5, and S1 can particularly affect the muscles in the lower extremities, including the plantar flexor muscles, which are crucial for movements like walking, running, and maintaining balance

ELIGIBILITY:
Inclusion Criteria:

* All patient diagnosed and referred from a physician
* Patients suffered from lumbar spondylosis (L4: L5) with radiculopathy more than 3 months
* Participants will be from both gender
* Age will be ranged from 30 to 50.
* BMI of all participants ≤ 30 kg/m2

Exclusion Criteria:

* Pregnant and breast-feeding women
* Patients diagnosed with depression and anxiety
* Patient who had undergone lumbar spine surgery
* People with systemic illnesses or physical deformities

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: one hundred thirty-two subjects (who have chronic lumbar spondylosis); from both genders will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
life disability | up to one day
  WHOQOL questionnaire will be used to assess life disability. it is defined as the individual's perception of their QoL. It consists of 24 questions which cover 4 categories plus 2 questions related to scale and health satisfaction. Each individual item of the WHOQOL-BRIEF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale.

SECONDARY OUTCOMES:
sciatic radiculopathy | up to one day
  The straight leg raise test will be used to assess lumbar radiclulopathy..The straight leg raise test is performed with the patient in a supine position. The examiner gently raises the patient's leg by flexing the hip with the knee in extension, and the test is considered positive when the patient experiences pain along the lower limb in the same distribution of the lower radicular nerve roots (usually L5 or S1).
  Furthermore, a positive straight leg raise test is determined when pain is elicited by lower limb flexion at an angle lower than 45 degrees. Patients usually request that the examiner abort the maneuver during the test if the pain is reproduced during the leg straightening. The buttock pain is usually relieved by flexing the patient's knee. Additional maneuvers have been described to enhance the test's sensitivity, such as the Bragaad sign, which consists of concomitant foot dorsiflexion to increase the pain while the examiner completes the leg raise
mechanosensitivity of the neuromeningeal structures within the vertebral canal | up to one day
  B. The Slump Test: is a neurodynamic test that is believed to evaluate the mechanosensitivity of the neuromeningeal structures within the vertebral canal.To perform the slump test, the patient is placed in an erect sitting position with the knees flexed to 90 and the legs hanging off of the side of the examination table The patient is asked to sit in a slouched position (thoracic and lumbar flexion with a posterior pelvic tilt) and is then requested to actively flex the cervical spine as far as comfortably possible. The clinician/physical therapist then applies gentle overpressure to the upper thoracic and lower cervical spine and maintains this position throughout the examination. The patient's ankle is then passively dorsiflexed to a neutral position while the knee is slowly passively extended until full extension is achieved